CLINICAL TRIAL: NCT05579522
Title: Clinical Evaluation of Interdental Papilla Reconstruction Using Injectable Autogenous Fat Compared To Hyaluronic Acid In Patients With Interdental Papillary Deficiency: A Randomized Controlled Clinical Trial.
Brief Title: Clinical Evaluation of Interdental Papilla Reconstruction Using Injectable Autogenous Fat Versus Hyaluronic Acid Filler.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal El Din Abd El Salam, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER313
Record Dates: First submitted 2022-10-07; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Hyaluronic Acid; Fat Graft
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- injectable fat graft (Experimental): Injection of fat graft from the buccal pad of fat into the interdental papilla
  Interventions: Procedure: Fat graft injection
- hyaluronic acid filler (Active Comparator): injection of hyaluronic acid filler in the interdental papilla
  Interventions: Procedure: Hyaluronic acid injection

INTERVENTIONS:
Procedure: Fat graft injection — Fat graft injection in the interdental papilla.
  Arms: injectable fat graft
Procedure: Hyaluronic acid injection — Hyaluronic acid injection in the interdental papilla
  Arms: hyaluronic acid filler

SUMMARY:
The goal of this randomized controlled trial is to evaluate the amount of interdental papilla fill following the injection of the fat graft compared to hyaluronic acid filler in patients with interdental papilla deficiency. Highly motivated patients having at least one deficient papilla with the presence of a contact point between adjacent teeth in the inter-bicuspid region. Papillary deficiency types I or II, according to Nordland and Tarnow (1998)classification will be selected. The main question it aims to answer is: In patient with interdental papillary deficiency, will injecting autogenous fat increase papilla height compared to hyaluronic acid injection? Participants in the test group will receive fat graft injection in the inter dental papilla. In the injection phase, 3 injections will be given at each papilla site: at baseline, 3 and 6 weeks intervals. While in the control group, hyaluronic acid injection in the interdental papilla and also 3 injections will be given at each papilla site at the same intervals.

DETAILED DESCRIPTION:
The treatment protocol will be divided into 3 phases: the pre-operative phase, where patients will be examined for eligibility, the treatment phase, where both control and interventional treatments will be carried out and finally the follow up phase, where patients will be followed up for the duration of the study.

A- Preoperative Evaluation A.1. Medical History A thorough detailed personal and dental history will be collected from all patients. Medical evaluation will be done before enrolling patients in the study to exclude the presence of any disease that may contraindicate treatment or exclude the patient from the study.

A.2. Clinical evaluation Initial periodontal therapy including full mouth supragingival scaling and subgingival debridement and patient motivation and education for proper oral hygiene.

After 6 weeks, re-evaluation of the deficient papilla will be done, and the degree of papillary deficiency according to Nordland and Tarnow classification [13] will be determined. Plaque and gingival indices will also be assessed and used to determine eligibility. Only patients with deficient papilla fulfilling the inclusion criteria will be recalled discussing all treatment options and sign the informed consent.

Once enrolled in the study, alginate impression will be taken for the involved arch/arches to construct study casts and fabricate customized stents to standardize measurements throughout the study. Standardized digital clinical photographs will also be taken for the GBT as a baseline measurement of the dimension of the black triangle. One-week later patients will be scheduled for the 1st injection.

A.3. Radiographic evaluation The distance between the contact area and inter-proximal bone crest (CP-BC) will then be measured to determine eligibility at the sites of papillary deficiency using peri-apical radiographs with paralleling technique and then confirmed by bone sounding.

B- Treatment phase:

In the injection phase, 3 injections will be given at each papilla site: at baseline, 3 and 6 weeks intervals.

1. Clinical measurement of the height of the black triangle will be by measuring the distance between the deficient papilla tip and contact area (PT-CP distance) to the nearest 0.5 mm (baseline). This will be done using a graduated periodontal probe and the fabricated customized stent for proper and standardized positioning of the probe at each measurement interval.
2. Standardized digital clinical photographs will be taken for the eligible deficient papillae for the baseline measurement of the surface area of black triangles.
3. Local anesthesia will be administered by infiltration to achieve the necessary anesthesia to allow a comfortable treatment procedure.
4. Patient allocation concealment will be broken to determine will treatment:

The patient will be randomly assigned to one of the treatment groups:

* Group A (Test): Fat graft injection in the inter dental papilla.
* Group B (Control): Hyaluronic acid injection in the interdental papilla.

Control group (Hyaluronic acid injection in the interdental papilla):

* The deficient papilla will be injected with 0.1 mm of HA gel concentration of 20 mg/ml using a 30-gauge disposable insulin syringe.
* The needle will be inserted 2-3 mm apical to the tip of the interdental papilla and directed coronally with an angulation of 45° to the long axis of the tooth, and the bevel directed apically.
* The papilla will be lightly molded in an incisal direction for 1 minute using gauze.

Test group (Fat graft injection in the inter dental papilla):

* Free buccal fat graft will be harvested from the buccal pad of fat.
* After administering anesthesia in the posterior area at the depth of the vestibule, a small horizontal incision in the free mucosa above the second and the third maxillary molars will be created using a sharp #11 blade.
* Through blunt dissection, the fat tissue will be accessed and easily mobilized into the oral cavity by progressive blunt dissection.
* The desired amount of fat will be harvested, and the remaining buccal pad will be pushed back in its place.
* Interrupted sutures with 5-0 vicryl resorbable sutures will be used to achieve primary closure of the incision.
* The fat graft will be rinsed to remove any debris and mechanically emulsified.

Fat emulsification

* Emulsiﬁcation of the fat will be done by shifting the fat between two 10-cc syringes connected to each other by a female-to-female Luer-Lok connector processing the block fat graft into nano-fat (Tonnard et al., 2013).
* After 30 passes, the fatty liquid will be ﬁltered over a sterile nylon cloth and the fluid will be collected in a sterile syringe. This is done to remove any connective tissue remnants that could block the ﬁne needles.
* A 30-gauge disposable insulin syringe will be used to load the nano-fat graft and will be inserted 2-3 mm apical to the tip of the interdental papilla.

Postoperative phase:

After completion of the treatment, self-care instruction will be given to the patients

Patient self-care instructions (Heitz-Mayfield 2008):

* Avoid mechanical plaque control in the area for 24 hours after the injection.
* Oral hygiene should be maintain using a soft toothbrush after the first 24 hours.
* Antiseptic mouth rinse, Chlorhexidine mouth rinse will be prescribed twice per day for two weeks.

Follow up and post-operative evaluation Patients will be recalled after 3 and 6 months from the first injection where clinical measurement of the gingival black triangle dimensions and standardized digital clinical photographs will be retaken.

The outcomes are:

1. Black triangle height

   * The black triangle height (BTH) will be assessed using standardized digital clinical photographs and analyzed by an image analysis program (Photoshop Cs 5, Adobe Systems, San Jose, CA, USA).
   * Method of aggregation: Mean
   * Specific measurement time point: at baseline, after 3 weeks, 6 weeks and 6 months postoperatively.
2. Black triangle area

   * The surface area of the black triangle (BTA) will be assessed using standardized digital clinical photographs and analyzed by an image analysis program (Photoshop Cs 5, Adobe Systems, San Jose, CA, USA).
   * Method of aggregation: Mean
   * Specific measurement time point: at baseline, after 3 weeks, 6 weeks and 6 months postoperatively.
3. Black triangle width

   * The black triangle width (BTW) will be assessed using standardized digital clinical photographs and analyzed by an image analysis program (Photoshop Cs 5, Adobe Systems, San Jose, CA, USA).
   * Method of aggregation: Mean
   * Specific measurement time point: at baseline, after 3 weeks, 6 weeks and 6 months postoperatively.
4. Post-Surgical Patient Satisfaction:

   * A 3-item questionnaire will be asked to the patients and a VAS scale for 0-10 will be used.
   * These items will be: Would you experience the same procedure another time? To what extent are you satisfied about the procedure? To what extent are you satisfied with the results?
5. Post-operative pain Visual Analogue Scale (VAS) with numbers from 0 to 10 ('no pain' to 'worst pain imaginable') will be measured at 24 hours.

Criteria for Discontinuing or Modifying Intervention:

Intervention will be discontinued or modified if the patient is unable to commit to the follow-up schedule or has any conditions that prevents him/her to continue the study.

Strategies to improve adherence to intervention:

* Patients will be recalled monthly for supportive periodontal therapy during the course of the study.
* Close follow up by phone will be done to ensure patient engagement

ELIGIBILITY:
Inclusion Criteria:

* Highly motivated patients having at least one deficient papilla in the inter-bicuspid region.
* Papillary deficiency types I or II, according to Nordland and Tarnow classification [13]
* No radiographic evidence of bone loss interproximally. (Cardaropoli et al,2004)
* Full mouth plaque index (PI) and gingival index (GI) scores should be less than 20%.
* No open contacts between affected teeth should be present.
* Teeth free from caries, proximal restorations, fixed prosthesis or orthodontic appliances

Exclusion Criteria:

* Subjects with medical conditions that may affect periodontal healing or regeneration.
* Subjects with a history of allergic reactions, smokers, and alcoholics
* Pregnant or breastfeeding females
* Patients with current or previous drugs intake that may predispose to gingival enlargement.
* Patients under orthodontic treatment or had orthodontic treatment in the past six months
* Patients with a history of periodontal surgeries over the last six months at the area of interest

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
change in Black Triangle Height (BTH) | Specific measurement time point: at baseline and after 6 months postoperatively.
  • The black triangle height (BTH) will be assessed using standardized digital clinical photographs and analyzed by an image analysis program (Photoshop Cs 5, Adobe Systems, San Jose, CA, USA).

SECONDARY OUTCOMES:
change in Black triangle area | Specific measurement time point: at baseline and after 6 months postoperatively.
  • The surface area of the black triangle (BTA) will be assessed using standardized digital clinical photographs and analyzed by an image analysis program (Photoshop Cs 5, Adobe Systems, San Jose, CA, USA).
change in Black triangle width | Specific measurement time point: at baseline and after 6 months postoperatively.
  The black triangle width (BTW) will be assessed using standardized digital clinical photographs and analyzed by an image analysis program (Photoshop Cs 5, Adobe Systems, San Jose, CA, USA).
Post-operative pain | will be measured at 24 hours.
  Visual Analogue Scale (VAS) with numbers from 0 to 10 ('no pain' to 'worst pain imaginable')
Post-Surgical Patient Satisfaction: | will be measured after 1 week
  A 3-item questionnaire will be asked to the patients and a VAS scale for 0-10 will be used.
  These items will be: Would you experience the same procedure another time? To what extent are you satisfied about the procedure? To what extent are you satisfied with the results?

IPD SHARING:
Plan to Share IPD: Undecided
the protocol, the results and the conclusion